CLINICAL TRIAL: NCT07162610
Title: A Multicenter, Randomized, Subject & Evaluator-blinded, Matched Pairs, Non-inferiority, Medical Device Pivotal Study to Evaluate the Efficacy and Safety of Injection With Rejuviel V® With Lidocaine as Compared to JUVEDERM® VOLUMA® With Lidocaine for Temporary Restoration of Mid-face Volume
Brief Title: Efficacy and Safety of Rejuviel V in the Correction of Midface Volume Deficit
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: PharmaResearch Co.,Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PR-Rejuviel-P3-01
Record Dates: First submitted 2025-08-31; First posted 2025-09-09 (Actual); Last update posted 2025-09-09 (Actual); Status verified 2025-08

CONDITIONS: Mid-face Volume Deficit
Keywords: Mid-face volume deficit; Mid face volume

STUDY DESIGN:
Intervention Model Description: Multicenter, Randomized, Subject & Evaluator-blinded, Matched Pairs, Non-inferiority
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Rejuviel V with lidocaine (Experimental): Single injection and optional touch up injection in Midface
  Interventions: Device: Rejuviel V® with lidocaine
- JUVEDERM® VOLUMA® with lidocaine (Active Comparator): Single injection and optional touch up injection in Midface
  Interventions: Device: JUVEDERM® VOLUMA® with lidocaine

INTERVENTIONS:
Device: Rejuviel V® with lidocaine — Crosslinked hyaluronic acid (HA) 22 mg/mL + 0.3% lidocaine hydrochloride.
  Other Names: Cleviel volume plus with lidocaine
  Arms: Rejuviel V with lidocaine
Device: JUVEDERM® VOLUMA® with lidocaine — Crosslinked hyaluronic acid (HA) 20 mg/mL + 0.3% lidocaine hydrochloride.
  Arms: JUVEDERM® VOLUMA® with lidocaine

SUMMARY:
The purpose is to evaluate the efficacy and confirm the safety of Rejeunesse Contour® with Lidocaine compared to Juvederm® Voluma® with Lidocaine for the temporary improvement of mid-face volume (including the cheekbone area, the anterior-medial cheek, and the area below the cheekbone).

The investigational medical device will be administered a total of once during the entire clinical trial period (or up to twice if additional treatment is required). After the administration, photographs of the application site and evaluations using the Mid-Face Volume Deficit Scale (MFVDS) will be conducted at 4 weeks, 12 weeks, 24 weeks, and 48 weeks. Satisfaction with mid-face volume improvement will be assessed using the Global Aesthetic Improvement Scale (GAIS). Additionally, changes in concomitant medications/treatments and adverse events will be reviewed in comparison to the previous visit.

ELIGIBILITY:
Inclusion Criteria:

* Korean men and women aged ≥30 years and ≤65 years at the time of informed consent.
* At screening, subjects with a score of 3 (moderate) or higher on the Mid Face Volume Deficit Scale (MFVDS), as assessed by independent on-site evaluators, with symmetrical deficits in both mid-face regions including the zygomatic area, anterior medial cheek, and subzygomatic area.
* Subjects who agree not to undergo any other procedures (e.g., filler injections other than the investigational medical device, laser treatment, chemical peeling, botulinum toxin, or facial plastic surgery) during the course of the clinical trial.
* Subjects who are able to understand and follow instructions and participate throughout the entire duration of the clinical trial.
* Subjects who voluntarily provide written informed consent to participate in the clinical trial.

Exclusion Criteria:

* History of anaphylaxis or severe allergic reactions requiring treatment.
* History of hypertrophic scars, keloids, or post-inflammatory hyperpigmentation.
* Use of anticoagulants (e.g., warfarin), antiplatelets, thrombolytics, immunosuppressants, or NSAIDs within 2 weeks prior to screening, or intake of other agents that may prolong coagulation time (e.g., vitamin E, garlic, ginkgo); Low-dose aspirin ≤300 mg/day permitted; participation allowed after ≥5 half-lives washout of the active compound.
* Use of topical facial medications (steroids, retinoids; excluding cosmetics) within 4 weeks prior to screening or planned during the study.
* Known hypersensitivity to investigational device components (sodium hyaluronate, lidocaine, lidocaine hydrochloride hydrate) or to amide-type local anesthetics (lidocaine, prilocaine, etc.).
* History of autoimmune disease (e.g., systemic lupus erythematosus, rheumatoid arthritis, autoimmune hepatitis, autoimmune hemolytic disease).
* History of sarcoidosis, granulomatous disease, or Osler's endocarditis.
* Active skin disease, inflammation, infection, scar, or wound at the treatment area.
* History or presence of herpetic eruption.
* Bleeding disorders.
* Severe hepatic dysfunction (ALT or AST >3 × ULN).
* Coagulation abnormalities (INR >1.5 × ULN).
* Prior or planned facial procedures/surgeries that may affect outcomes; permanent implants (e.g., PMMA, silicone, Gore-Tex) in treatment area.
* History of malignancy within the past 5 years.
* Drug or alcohol abuse.
* Heavy smoking (>20 cigarettes/day).
* Requirement for continuous immunosuppressive therapy during the study.
* Active inflammatory conditions requiring systemic anti-inflammatory treatment (including streptococcal diseases).
* Thin skin in the mid-face or fluid retention tendency in lower eyelids/infraorbital fat pads.
* Use of wrinkle-preventive medical devices or drugs in the mid-face within 3 months prior to screening, or planned during the study.
* Untreated epilepsy.
* Porphyria.
* Use of another investigational medical device or drug within 3 months prior to screening.
* Female subjects of childbearing potential who are unwilling to use medically acceptable contraception during the study, or who are pregnant, breastfeeding, or planning pregnancy.

Ages: 30 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 89 (Actual)
Dates: Start 2024-04-07 (Actual); Primary Completion 2026-03-08 (Estimated); Study Completion 2026-03-30 (Estimated)

PRIMARY OUTCOMES:
Percentage improvement in mid-face volume | at Weeks 24 after the final administration
  Percentage improvement in mid-face volume at Weeks 24 after the final administration of the investigational medical device, as assessed by independent photo evaluators compared with baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Chung-Ang University Hospital, Soeul, South Korea

IPD SHARING:
Plan to Share IPD: No